CLINICAL TRIAL: NCT05893576
Title: A Relative Bioavailability Study of Single-dose, Randomized, Open-label, Single-period, Parallel Design of HRS9531 Injection Using Different Manufacturing Processes in Healthy Subjects
Brief Title: A Relative Bioavailability Study of HRS9531 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-103
Record Dates: First submitted 2023-05-05; First posted 2023-06-08 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a single-dose, parallel design trial, consisting of two parallel groups: a reference formulation group (R: original formulation) and a test formulation group (T: new formulation). Both R and T groups receive a same dose of HRS9531.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R group (reference formulation group) (Experimental)
  Interventions: Drug: HRS9531
- T group (test formulation group) (Experimental)
  Interventions: Drug: HRS9531

INTERVENTIONS:
Drug: HRS9531 — Receive a single dose of HRS9531 of original formulation.
  Arms: R group (reference formulation group)
Drug: HRS9531 — Receive a single dose of HRS9531 of new formulation.
  Arms: T group (test formulation group)

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of the new formulation of HRS9531 injection between the original formulation of HRS9531 injection.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, be able and willing to provide a written informed consent;
2. Age 18-45 years on the date of signing informed consent (inclusive);
3. Body weight ≥50 kg for male and 45 kg for female, body mass index (BMI) within the range of 19.0-26.0 kg/m2 (inclusive);
4. Subjects with good general health, no clinically significant abnormalities.

Exclusion Criteria:

1. With previous major organ diseases, including but not limited to neuropsychiatric, cardiovascular, digestive, respiratory, urinary, endocrine, blood, immune and other diseases, are judged by researchers to be unsuitable for the study;
2. Had a severe trauma or major surgery within 6 months prior to screening, planned to undergo surgery during the trial period;
3. Participants in clinical trials of any drug or medical device in the 3 months prior to screening;
4. Blood donation history or blood loss ≥400 mL within 3 month or ≥200 mL within 1 month before screening, or received blood transfusion within 3 months;
5. Allergic constitution includes severe drug allergy or history of drug allergy;
6. Hepatitis B surface antigen (HBsAg), HIV antibody detection, hepatitis C virus antibody (HCVAb), treponema pallidum specific antibody detection, positive;
7. Breast-feeding women;
8. The investigator considers that the subject has any other factors that would make it inappropriate to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration versus time curve (AUC) of HRS953 | Start of treatment up to Day 43
Maximum Concentration (Cmax) of HRS9531 | Start of Treatment up to Day 43
Calculate the ratio of bioavailability between the new formulation and original formulation of HRS9531 according to the equation F (relative bioavailability) =AUCT·DR/AUCR·DT×100% | Start of Treatment up to Day 43

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | Start of Treatment up to Day 43
Apparent terminal half-life (t1/2) | Start of Treatment up to Day 43
Clearance (CL/F) | Start of Treatment up to Day 43
Apparent volume of distribution (VzF) | Start of Treatment up to Day 43
Incidence and severity of adverse events | Screening period up to Day 43

CONTACTS AND LOCATIONS:
Locations (1):
- Central hospital affiliated to Shandong first mecical university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided